CLINICAL TRIAL: NCT04446299
Title: A Safety and Efficacy Comparison of BLI4900 Bowel Preparation Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Brief Title: Study 301: BLI4900 Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI4900-301
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLI4900 (Experimental): Experimental bowel preparation solution for oral ingestion
  Interventions: Drug: Bowel Prep
- FDA Approved Control (Active Comparator): FDA approved bowel preparation solution for oral ingestion
  Interventions: Drug: Bowel Prep

INTERVENTIONS:
Drug: Bowel Prep — Orally ingested liquid bowel preparation

SUMMARY:
The purpose of this study is to compare the safety and efficacy of BLI4900 bowel preparation to an FDA-approved control as 2-day, split-dose bowel preparations prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* 18 to 85 years of age (inclusive)
* If female, and of child-bearing potential, is using an acceptable form of birth control.
* Negative serum pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastroparesis, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects with inflammatory bowel disease who have a history of any bowel resection (small intestine or colon), suspected active inflammation, or symptoms suggestive of obstruction or known bowel stricture.
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects who have regularly used laxatives or colon motility altering drugs in the last month (i.e. more than 2-3 times per week) and/or laxative use within 72 hours prior to administration of the preparation
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
* Subjects taking diuretics, anti-hypertensive medications, including angiotensin converting enzyme (ACE) inhibitors and Angiotensin II receptor blockers (ARBs), or chronic NSAIDs, that have not been stable for 30 days.
* Subjects with uncontrolled hypertension.
* Subjects taking antibiotics within 7 days of colonoscopy.
* Subjects with severe renal, hepatic or cardiac insufficiency.
* Subjects with an abnormal and clinically significant physical examination or ECG finding at Visit 1.
* Subjects undergoing insulin therapy for any indication.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.
* Subjects taking tricyclic antidepressants.
* Subjects using drugs of abuse, including abused prescription medications.
* Subjects who are withdrawing from alcohol or benzodiazepines.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories / Sebela Pharmaceuticals
Locations (25):
- United States (25):
  - 301 Research Site 18, Huntsville, Alabama
  - 301 Research Site 24, Sun City, Arizona
  - 301 Research Site 7, San Diego, California
  - 301 Research Site 16, Clearwater, Florida
  - 301 Research Site 12, Jacksonville, Florida
  - 301 Research Site 9, Palm Harbor, Florida
  - 301 Research Site 4, Palmetto Bay, Florida
  - 301 Research Site 26, Port Orange, Florida
  - 301 Research Site 14, St. Petersburg, Florida
  - 301 Research Site 25, Sunrise, Florida
  - 301 Research Site 2, Decatur, Georgia
  - 301 Research Site 10, Indianapolis, Indiana
  - 301 Research Site 3, Monroe, Louisiana
  - 301 Research Site 17, Shreveport, Louisiana
  - 301 Research Site 11, Flowood, Mississippi
  - 301 Research Site 13, Chesterfield, Missouri
  - 301 Research Site 19, Reno, Nevada
  - 301 Research Site 15, Brooklyn, New York
  - 301 Research Site 5, Great Neck, New York
  - 301 Research Site 23, New York, New York
  - 301 Research Site 6, Raleigh, North Carolina
  - 301 Research Site 21, Mentor, Ohio
  - 301 Research Site 20, Hixson, Tennessee
  - 301 Research Site 1, Ogden, Utah
  - 301 Research Site 22, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI4900 | FDA Approved Control
Started | 259 | 260
Completed | 220 | 230
Not Completed | 39 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI4900 | FDA Approved Control | Total
Number analyzed (Participants) | 259 | 260 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.4) | 57.3 (11.5) | 56.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 148 | 283
  Male | 124 | 112 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 18 | 39
  Not Hispanic or Latino | 238 | 241 | 479
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 73 | 69 | 142
  White | 175 | 182 | 357
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 259 | 260 | 519

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Successful Bowel Preparation
Description: Successful bowel preparation is defined as a preparation rated as Excellent or Good by the blinded endoscopist on a 4 point scale (Excellent, Good, Fair, Poor).
Time Frame: 2 days
Population: Modified intent-to-treat population - subjects who took any portion of the study preparation and did not discontinue due to a reason other than safety, efficacy or tolerability.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4900 | FDA Approved Control
Number analyzed (Participants) | 232 | 239
Participants | 215 | 212
Statistical Analysis 1: Comparison: BLI4900 vs FDA Approved Control; Test type: Non-Inferiority — The predetermined non-inferiority margin was 10%; p < 0.001, Mantel Haenszel; Risk Difference (RD) = 3.42, 95% CI 2-sided [-1.68 to 8.52]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The Analysis Population for adverse event reporting, including serious adverse events and all cause mortality, is the Safety Population which includes all patients that took any portion of the study preparation. This population differs from the Baseline Population because some patients that were dispensed a study preparation did not take it.
Arm/Group | BLI4900 | FDA Approved Control
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/243
Serious Adverse Events (participants affected / at risk) | 1/233 | 0/243
Other Adverse Events (participants affected / at risk) | 46/233 | 34/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI4900 (N=233) | FDA Approved Control (N=243)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4900 (N=233) | FDA Approved Control (N=243)
Nausea (Gastrointestinal disorders) | 30 | 22
Abdominal distension (Gastrointestinal disorders) | 14 | 6
Vomiting (Gastrointestinal disorders) | 13 | 7
Abdominal Pain (Gastrointestinal disorders) | 7 | 9
Headache (Nervous system disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04446299/Prot_SAP_000.pdf